CLINICAL TRIAL: NCT05109338
Title: Efficacy of Ben-Guard Garment in Reducing the Frequency of Pediatric Central Line Complications: A Pilot Study
Brief Title: Efficacy of Ben-Guard Garment in Reducing Pediatric Central Line Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-0781; Protocol Version 8/3/2021 (Other: UW Madison); A539790 (Other: UW Madison); fund for garments (Other Grant/Funding Number: Cars Curing Kids)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Central Venous Catheters
Keywords: Central venous catheter; complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ben-Guard user (Experimental): Participants will wear the garment for up to 18 months while needing a central line catheter.
  Interventions: Device: Ben-Guard Garment
- Retrospective match control (No Intervention): Matched historical control for intervention group based on age, gender and duration of use of a central venous catheter.

INTERVENTIONS:
Device: Ben-Guard Garment — Wearable device designed to secure CVCs and gastrointestinal feeding tubes. The Ben-Guard Catheter Securement Device was designed specifically to better secure and conceal CVC tubing, protecting the patient by keeping tubing closer to the body.
  Arms: Ben-Guard user

SUMMARY:
Central venous catheter (CVC) insertion is a common surgical procedure performed in children for the delivery of nutritional support, medications, frequent blood draws or transfusions. Maintaining hygienic conditions is absolutely necessary in order to avoid contamination of the catheter and tubing to avoid bloodstream infections. Fractures in the tubing is a common complication that places children at increased risk for infections. In order to help keep the tubing stable to avoid fractures and dislodgements, a wearable device was created called Ben-Guard. This pilot study is being undertaken to determine if the Ben-Guard device will reduce the incidence and severity of adverse events in children requiring CVCs.

DETAILED DESCRIPTION:
Conduct a pragmatic pilot study of the Ben-Guard Catheter Safety Device in 40 pediatric patients with central venous catheters (CVC). Participants will be issued 3-5 garments, which are expected to be worn at all times. This study will be conducted over an 18 month period. Participants are expected to wear the garment daily for the duration of the study (or duration of their treatment if <18 months). Data will be reviewed every 3 months to measure the garment's acceptability and effect on the frequency of central line-associated complications. Outcomes will be compared to a matched retrospective cohort. This study will use the device consistent with the description as a registered FDA Class 1 device. The investigators are conducting this study to clinically and scientifically evaluate the device's ability to change the frequency of CVC fractures and CVC complications in children.

ELIGIBILITY:
Inclusion Criteria:

* Participants age 0-10
* medical disease or condition that requires a CVC for treatment, supportive care or nutritional support
* English Speaking

Exclusion Criteria:

* Any patient who received a non-tunneled CVC
* Any patient who had a tunneled CVC placed from an outside institution
* Age > 10
* Patients that cannot communicate or read English

Ages: 0 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Mean Number of CVC Fractures | Up to 18 months
  compared to retrospective cohort

SECONDARY OUTCOMES:
Mean Number of CVC Dislodgements | Up to 18 months
  The frequency of CVC dislodgements compared to a matched retrospective cohort.
Total Number of Central-Line Associated Blood Stream Infections (CLABSIs) | Up to 18 months
  Number of central-line associated blood stream infections compared to a matched retrospective cohort.
Total Number of CVC-related Emergency Department or Urgent Care Visits | Up to 18 months
  The number of CVC-related emergency department visits compared to a matched retrospective cohort.
Mean CVC-related Total Healthcare Associated Costs | Up to 18 months
  Mean CVC-related total healthcare-associated costs compared to a matched retrospective cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nichol, MD, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- American Family Children's Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No